CLINICAL TRIAL: NCT03755375
Title: The Effects of Physiotherapeutic Interventions Applied to the Bladder Pain Syndrome: A Randomized Control Trial
Brief Title: Physiotherapeutic Interventions Applied to the Bladder Pain Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Responsible Party: Principal Investigator, Clarice Tanaka, PhD, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 61595016.0.0000.0068
Record Dates: First submitted 2018-10-11; First posted 2018-11-28 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Interstitial Cystitis; Painful Bladder Syndrome; Bladder Pain Syndrome
Keywords: Bladder pain syndrome; Physical therapy; Postural balance; Manual therapy; Biofeedback
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Transcutaneous Electric Nerve Stimulation; Biofeedback, Psychology; Musculoskeletal Manipulations

STUDY DESIGN:
Intervention Model Description: Randomized control trial. All patients will be randomized by the computer (www.random.org) in 3 groups of treatment. Then, they were assessed by specialized physiotherapists through a medical history data; application of validated questionnaires of pain, urinary symptoms, sexual function and quality of life; pelvic floor muscles physical and surface electromyographic assessment. Patients were randomized to 3 different treatment groups, and treatment consisted by 10 sessions, once a week. TENS group was treated using Biofeedback , manual therapy and transcutaneous electrostimulation. Postural group was treated using Biofeedback , manual therapy and postural exercises. Conventional group was treated using Biofeedback and manual therapy. All participants were evaluated post treatment and at 3 months of follow-up using the same procedures of the initial assessment.
Who Masked: Participant
Masking Description: After the assessment, participants were blinded randomized by a mask researcher using random.org and allocated into three groups of treatment (TENS, Postural and Conventional) held over 10 sessions once a week.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- E-stim Group (Active Comparator): TENS group was treated with biofeedback, manual therapy, andtranscutaneous electrostimulation (TENS), a peripheral neuromodulation to promote analgesia in pain areas, using two transcutaneous self-adhesive electrodes Axelgaard 5 cm x 5 cm with 2 cm of distance between them. The parameters used were frequency = 100 Hz, pulse width = 50-100 µs, and current intensity according to the patient's sensitivity.
  Interventions: Device: TENS; Device: Biofeedback; Behavioral: Manual therapy
- Postural Group (Active Comparator): Postural group was treated with biofeedback, manual therapy, and postural exercises , which promoted pelvic mobility and functional training associated with respiratory exercises increasing the diaphragmatic excursion.Postural exercises consisted of 10 repetitions of breathing exercises in the lay-down position, 10 repetitions of hip anteversion and retroversion in the sitting position, and 10 repetitions of hip anteversion, retroversion, and lateral movement in the stand-up position.
  Interventions: Behavioral: Postural exercises; Device: Biofeedback; Behavioral: Manual therapy
- Conventional Group (Active Comparator): Conventional group was treated with biofeedback for pelvic floor relaxation and manual therapy to release the tension in the suprapubic, pelvic, and intravaginal areas. The manual therapy consisted of a myofascial trigger point release maneuver using digital pressure and muscle fiber stretching in pain areas. Biofeedback consisted of pelvic floor muscle coordination and relaxation exercises using intravaginal probes. The training program was initiated with 10 fast contractions with 5 seconds of relaxation between them followed by 10 sustained contractions of 5 seconds with 10 seconds of relaxation between them. Finally, one minute of pelvic floor relaxation was performed.
  Interventions: Device: Biofeedback; Behavioral: Manual therapy

INTERVENTIONS:
Device: TENS — transcutaneous electrostimulation to improve the pain.
  Arms: E-stim Group
Behavioral: Postural exercises — breathing exercises in the lay-down position, hip anteversion and retroversion in the sitting position, and anteversion, retroversion, and lateral movement in the stand-up position
  Arms: Postural Group
Device: Biofeedback — pelvic floor muscle coordination and relaxation exercises using intravaginal probes
Behavioral: Manual therapy — myofascial trigger point release maneuver using digital pressure and muscle fiber stretching in pain areas

SUMMARY:
Related to urological and gynecological systems, patients with Bladdeer Pain Syndrome (BPS) often present pain, pressure and chronic discomfort in suprapubic and perineal area associated with low urinary tract symptoms. This condition can generates a negative impact in cognitive, social, behavioral and sexual quality of life.

As Bladder Pain Syndrome originates from different causes and includes the genitourinary, gastrointestinal, musculoskeletal and neuropsychological systems, a multidisciplinary approach is needed with doctors,physiotherapists, psychologists and others. Physiotherapeutic interventions are recommended as a conservative treatment for patients with BPS. The physiotherapeutic interventions include the use of Biofeedback to relax the pelvic floor muscles and manual therapy (myofascial trigger points release) to decrease muscle tension. Transcutaneous electrostimulation (TENS) is used to decrease the pain and postural exercises to improve the pelvic mobility. In this study, our hypothesis was that women with BPS presented musculoskeletal dysfunction, and we tested a different physiotherapy approach that was not being used. The reason for that understanding was the presence of refractory urinary and pain symptoms notwithstanding the physiotherapy conventional treatment, such as manual therapy and biofeedback. To test our hypothesis, we decided to add either TENS or postural exercises to the conventional treatment. The objective of this study was to verify the effects of biofeedback (BF) and manual therapy (MT) associated with transcutaneous electrical nerve stimulation (TENS) or postural exercises (PE) in the treatment of bladder pain syndrome (BPS) in women regarding pain and urinary symptoms.

DETAILED DESCRIPTION:
In the initial assessment, two specialized and trained physiotherapists applied a demographic questionnaire to identify the characteristics of the sample and validated questionnaires of perineal and suprapubic pain (Visual Analog Scale of Pain [VAS])(21) to quantify the pain; urinary symptoms and problems (O'Leary-Sant - The Interstitial Cystitis Symptom and Problem Index) (22) to evaluate the presence of urgency, frequency, nocturia and to quantify how much these symptoms represent a problem to the patients, and the Female Sexual Function Index (FSFI) (23) to evaluate the impact on sexual life. Then, a physical assessment by the inspection and palpation of pelvic and perineal areas was made to identify myofascial trigger points.

After the assessment, participants were blinded randomized by a mask researcher using random.org and allocated into three groups of treatment (TENS, Postural and Conventional) held over 10 sessions once a week. All participants needed to attend the whole treatment to be included with a maximum delay of 2 weeks to start treatment. Conventional group was treated with biofeedback for pelvic floor relaxation and manual therapy to release the tension in the suprapubic, pelvic, and intravaginal areas. The manual therapy consisted of a myofascial trigger point release maneuver using digital pressure and muscle fiber stretching in pain areas. Biofeedback consisted of pelvic floor muscle coordination and relaxation exercises using intravaginal probes. The training program was initiated with 10 fast contractions with 5 seconds of relaxation between them followed by 10 sustained contractions of 5 seconds with 10 seconds of relaxation between them. Finally, one minute of pelvic floor relaxation was performed.

TENS group was treated with biofeedback, manual therapy, and transcutaneous electrostimulation (TENS), a peripheral neuromodulation to promote analgesia in pain areas, using two transcutaneous self-adhesive electrodes Axelgaard 5 cm x 5 cm with 2 cm of distance between them. The parameters used were frequency = 100 Hz, pulse width = 50-100 µs, and current intensity according to the patient's sensitivity.

Postural group was treated with biofeedback, manual therapy, and postural exercises , which promoted pelvic mobility and functional training associated with respiratory exercises increasing the diaphragmatic excursion. Postural exercises consisted of 10 repetitions of breathing exercises in the lay-down position, 10 repetitions of hip anteversion and retroversion in the sitting position, and 10 repetitions of hip anteversion, retroversion, and lateral movement in the stand-up position.

The biofeedback and TENS device used was a Myotrac Infiniti T9800 (Thought Technology Ltda., Montreal, Canada, ISO 13485:2016ISO 13485:2016), a 2-channel system of surface electromyography and electrostimulation using the Biograph Infiniti platform. For biofeedback training, we used intravaginal electrodes St-Cloud/Femelex 6.9 cm.

All participants were evaluated post treatment and at 3 months of follow-up using the same procedures of the initial assessment.

All participants were instructed to perform home training daily 3 times/day during treatment and completed an exercise diary to demonstrate adherence to treatment. TENS and Conventional groups were instructed to perform pelvic floor relaxation exercises, and Postural group was instructed to perform pelvic floor relaxation exercises plus postural exercises.

ELIGIBILITY:
Inclusion criteria: women with a diagnosis of BPS according to NIH clinical criteria ≥ 18 years old, who presented symptoms of perineal and suprapubic pain, using painkillers, anticholinergics, antidepressants, and anticonvulsants for at least 6 months, and exhibited absence of urinary infection for at least 3 months for the initial assessment.

Exclusion criteria: women with positive uroculture, under actual or previous oncologic treatment, with systemic or neurological diseases that could compromise pelvic structures, with cognitive deficiency that compromised the understanding of the provided instructions and those who refused to participate in the study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2019-12-19 (Actual); Study Completion 2019-12-19 (Actual)

PRIMARY OUTCOMES:
Pain symptoms | up to 3 months
  Change from Baseline in pain sympotms on the Visual Analog Scale after treatment
Urinary symptoms | up to 3 months
  Change from Baseline in urinary symptoms on the O'Leary- Sant Urinary symptoms and problems score after treatment

SECONDARY OUTCOMES:
Sexual activity | up to 3 months
  Change from Baseline in Female sexual function index score after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Clarice Tanaka, PhD, Study Director — University of Sao Paulo; Homero Bruschini, PhD, Study Chair — University of Sao Paulo
Locations (1):
- Universidade de São Paulo, São Paulo, Brazil